CLINICAL TRIAL: NCT05966987
Title: Assessment of Different Orthodontic Tooth Movements Assisted With Low-level Laser Therapy vs. Injectable Plasma-rich Fibrin: A Comparative Clinical Investigation
Brief Title: Assessment of Different Orthodontic Tooth Movements Assisted With Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 923/91
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Injectable Plasma-rich Fibrin Versus Low-Level Laser Therapy on Othodontic Movement

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- i-PRF side: canine retraction (Experimental): application of i-PRF with translation of maxillary canine that will be performed on intervention sides according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- i-prf side control side (No Intervention): i-PRF side:canine retraction control side
- LLLT side canine retraction (Experimental): translation of maxillary canine that will be performed with LLLT application according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- LLLT side canine retraction control side (No Intervention): LLLT side canine retraction control side wihout intervention
- I-PRF groupMolar distalization group inrervention side (Experimental): Idistalization assisted with Injectable platelet-rich fibrin (i-PRF) according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- I-PRF groupMolar distalization group control side (No Intervention): distalization without i-PRF intervention
- LLLT group: distalization intervntion side (Experimental): distalization will be commenced with application of LLLT according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- LLLT group: distalization control side (No Intervention): distalization will be commenced without application of LLLT according to a standardized protocol
- i-PRF group: leveling and alignment (Experimental): leveling and alignment assisted with Injectable platelet-rich fibrin (i-PRF) according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- LLLT group: leveling and alignment (Experimental): leveling and alignment be commenced with application of LLLT according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- leveling and alignment without intervention (No Intervention): leveling and alignment without intervention
- I-PRF group: Intrusion (Experimental): intrusion assisted with Injectable platelet-rich fibrin (i-PRF) according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- LLLT group: Intrusion (Experimental): intrusion assisted with application of LLLT according to a standardized protocol
  Interventions: Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin
- intrusion control group (No Intervention): intrusion without intervention

INTERVENTIONS:
Combination Product: Low-level Laser Therapy vs. Injectable Platelets-rich Fibrin — laser and platelet rich fibrin
  Arms: I-PRF group: Intrusion; I-PRF groupMolar distalization group inrervention side; LLLT group: Intrusion; LLLT group: distalization intervntion side; LLLT group: leveling and alignment; LLLT side canine retraction; i-PRF group: leveling and alignment; i-PRF side: canine retraction

SUMMARY:
The present prospective clinical study will be undertaken for assessment of the effect of application of Injectable plasma-rich fibrin versus Low-Level Laser Therapy onthe rate of different orthodontic tooth movements,

DETAILED DESCRIPTION:
The present prospective clinical study will be undertaken for assessment of the effect of application of Inject able plasma-rich fibrin versus Low-Level Laser Therapy on the rate of different orthodontic tooth movements, namely: canine retraction, mandibular incisors leveling and alignment, maxillary molar distalization and maxillary incisor intrusion.

ELIGIBILITY:
Inclusion Criteria:

A- leveling and alignment Eligibility criteria

1. Complete permanent dentition (third molars not included).
2. Moderate mandibular anterior crowding (with Little's irregularity index score greater than 4 mm) who required nonextraction approach in the mandibular arch.
3. No tooth size, shape or root abnormalities visible on patient's radiographic records.
4. No spaces in the mandibular arch.
5. No blocked out tooth that did not allow for placement of the bracket at the initial bonding appointment.
6. No required management with interproximal stripping, intermaxillary elastics, open NiTi springs, and removable or extra-oral devices. Maxillary molar distalization Inclusion criteria:

1. Age ranges from 14 to 17 years. 2. Bilateral Class II molar relationship. 3. Skeletal Class I or mild Class II relationship. 4. Normal or decreased vertical height. 5. No posterior crowding or spaces. 6. Fully erupted maxillary first and second molars. 7. Congenitally missing or extracted third molars. 8. Good oral hygiene. 9. Absence of any periodontal disease and alveolar bone loss. 10. Absence of medications that may inhibit orthodontic movement

* Lower incisor leveling and alignment Inclusion criteria

  1. Complete permanent dentition (third molars not included);
  2. Moderate mandibular anterior crowding (with little's irregularity index score greater than 4 mm) who required non-extraction approach in the mandibular arch;
  3. No tooth size, shape or root abnormalities visible on the patient's radiographic records;
  4. No spaces in the mandibular arch;
  5. No blocked out tooth that did not allow for placement of the bracket at the

initial bonding appointment; 6. No required management with interproximal stripping, inter-maxillary elastics, open NiTi springs, and removable or extra-oral devices. Canine retraction Eligibility criteria

1. Age, 15 to 25 years;
2. Class ii division 1 malocclusion with mild or no crowding;
3. No previous orthodontic treatment;
4. No systemic disease that might have affected bone formation or density, such as osteoporosis, hyperparathyroidism, or vitamin d deficiency;
5. Adequate oral hygiene;
6. Probing depth values not exceeding 3 mm across the
7. Entire dentition;
8. Adequate thickness of the attached gingiva (1-2 mm);
9. No radiographic evidence of bone loss

Exclusion Criteria:Exclusion criteria:

1. Patients who required surgery to correct skeletal discrepancies.
2. Patients with congenital dentoskeletal disorders.
3. Missed or mutilated teeth in maxillary arch.
4. Patients with poor oral hygiene and/or periodontally compromised patients Severe dental crowding that necessitates an extraction approach 2. Abnormal anteroposterior and vertical relationships; 3. Patients with cleft lip and palate, anomalies, and syndromes; 4. Previous orthodontic 5. Treatment; 6. Regular medications intake that could interfere with otm. -

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
assessment of the effect of application of Injectable plasma-rich fibrin versus Low-Level Laser Therapy on the accelration rate of different orthodontic tooth movements by millimeter | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326
- [Result] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391